CLINICAL TRIAL: NCT03609736
Title: PSMA-based 18F-DCFPyL PET/CT: Evaluating Its Application in Real Life
Acronym: PEARL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Grand River Hospital (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Other Study IDs: PEARL
Record Dates: First submitted 2018-07-25; First posted 2018-08-01 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 18F-DCFPyL PET/CT — * A bolus of less than or equal to 9 mCi (333 MBq) of 18F-DCFPyL will be injected IV by slow IV push.
  * After administration of the 18F-DCFPyL the line will be flushed with saline (0.9% w/v).
  * Subjects should be encouraged to drink up to 500 mL of water shortly after the administration of 18F-DCFPyL.
  * At 60-minutes (± 10 minutes) after administration of 18F-DCFPyL, the PET/CT scan will be acquired with the subject in the supine position and the FOV including the mid-thighs to skull base.

SUMMARY:
The purpose of the study is to provide pilot data on the clinical situations in which ordering a 18F-DCFPyL positron emission tomography/computed tomography (PET/CT) was thought to be clinically useful, and to document how the results of the 18F-DCFPyL PET/CT affected patient management. The results of this study could then serve as a guide to help OHIP to consider these scenarios when deciding the precise indications for funded 18F-DCFPyL PET/CT scans in the future. In this study the investigators will image subjects with prostate cancer using 18F-DCFPyL PET/CT and record how the result of the study affected patient management.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Age ≥ 18 years and male
* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* One of the following:
* CT scan showing indeterminate lymph node(s) in the pelvis that could potentially be treated radically with radiotherapy if found to be positive on PSMA PET.
* Suspected oligometastatic disease (< 4 sites of disease) that could potentially be treated with stereotactic/radical doses of radiotherapy.

Exclusion Criteria:

* Serious or uncontrolled co-existent non-malignant disease, including active and uncontrolled infection
* Uncontrolled hypertension (systolic BP ≥ 160 mmHg or diastolic BP ≥ 95 mmHg)
* Condition or situation which, in the investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with subject's participation in the study
* Not willing to comply with the procedural requirements of this protocol
* Subjects who have partners of childbearing potential who are not willing to use a method of birth control with adequate barrier protection as determined to be acceptable by the principal investigator and sponsor during the study and for 13 weeks after last study drug administration.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate Cancer Patients
Study Population: This study will image male subjects with PCa using 18F-DCFPyL PET/CT for detection of disease with correlation to standard-of-care imaging (CT and bone scan) and clinical follow-up over a 1-year time period.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2018-08-10 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
To acquire pilot data on the use of 18F-DCFPyL PET/CT following conventional imaging (CT and bone scan) for the detection of metastases in men with prostate cancer | 1 year
  To acquire pilot data on the use of 18F-DCFPyL PET/CT following conventional imaging (CT and bone scan) for the detection of metastases in men with prostate cancer when: 1. The CT scan shows indeterminate lymph node(s) in the pelvis that could potentially be treated radically with radiotherapy if found to be positive on 18F-DCFPyL PET/CT; 2. The subject is suspected to have oligometastatic disease (< 4 sites of disease) that could potentially be treated with stereotactic/ radical doses of radiotherapy.

SECONDARY OUTCOMES:
To acquire pilot data comparing the number and location of metastatic lesions on 18F-DCFPyL PET/CT with standard of care imaging (CT and bone scan). | 1 year
To acquire pilot data on the change in management plans resulting from 18F-DCFPyL PET/CT compared with standard of care imaging (CT and bone scan). | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Grand River Hospital, Kitchener, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No